CLINICAL TRIAL: NCT06838052
Title: The Effect of Laughter Yoga-Supported Strong Woman, Safe Life Training Program on Attitudes Towards Violence, Styles of Coping with Stress and Psychological Flexibility
Acronym: Laughter Yoga
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Fatma Ozlem Ozturk, Assoc. Prof. Dr., Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AnkaraUnivesirtyNF
Record Dates: First submitted 2025-02-13; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Violence Against Women (VAW); Laughter Yoga; Intimate Partner Violence (IPV); Coping Skills; Resilience
Keywords: Woman, Married Persons, Laughter Yoga, Intimate partner violence, Stress,Coping Skills, Elasticity, Psychological, Resilience

STUDY DESIGN:
Intervention Model Description: The research will be conducted as a randomized controlled parallel group intervention study. The universe of the study will consist of 7988 women registered to 24 Women's Education and Culture Centers (KEKM) affiliated to Altındağ Municipality. 1 center will be randomly selected from 24 Women's Education and Culture Centers for the sample of the study. In this study, the smallest sample size was determined as 43 for each group, a total of 86, with 80% statistical power and α=.05 significance level. Considering 10% data loss in the determined sample size, it was planned to include a total of 94 participants, 47 for each group. The women included in the study will be assigned to the intervention (47 participants) and control (47 participants) groups by randomization. It is aimed to apply the Strong Woman, Safe Life Education Program Supported by Laughter Yoga to the participants in the intervention group face-to-face for an 8-week period. The 47 participants in the intervention group wil
Who Masked: Outcomes Assessor
Masking Description: The data will be evaluated by an independent statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The group where the Laughter Yoga-Strong Woman, Safe Life Training Program will be implemented (Experimental): Within the scope of the Laughter Yoga Supported Strong Woman, Safe Life Training Program, it is planned to provide 8 weeks of training to the participants in the intervention group.
  Interventions: Other: Strong Woman, Safe Life Training Program Supported by Laughter Yoga
- Control Group (No Intervention)

INTERVENTIONS:
Other: Strong Woman, Safe Life Training Program Supported by Laughter Yoga — The training program consists of 8 modules, each module consists of two sessions. A session will last 45 minutes. The program includes the following topics: Self-Awareness and Importance of Communication (Module 1), Stress and Coping Techniques (Module 2), Gender (Module 3), Women's Empowerment (Module 4), Violence and Its Effects on Women's Health (Module 5), Non-Violent Communication (Module 6), Combating Violence (Module 7), Psychological Health (Module 8). In addition, a laughter yoga session will be held in the second session of each module.
  Arms: The group where the Laughter Yoga-Strong Woman, Safe Life Training Program will be implemented

SUMMARY:
The aim of this project is to examine the effects of the Laughter Yoga Supported Strong Woman, Safe Life Education Program applied to women on attitudes towards violence, stress coping styles and psychological flexibility.

The problem of violence against women is a public health problem that affects and concerns not only women at the individual level, but also children, all family members and therefore society. According to the data of the Turkish Statistical Institute in our country, 38% of women have been subjected to spousal or partner violence at some point in their lives. Violence or the threat of violence that causes fear, pain and anxiety in women from an individual perspective; constitutes an obstacle to women's more active and productive participation in economic and social life, especially in the private sphere. From a social perspective, the economic cost of violence against women is extremely high in terms of loss of working hours and wages, social services, legal and medical expenses.

Our country has a culturally patriarchal social structure. Living in a patriarchal order affects beliefs and attitudes towards the acceptance of violence, making women more vulnerable to violence. Living in a patriarchal order affects beliefs and attitudes towards acceptance of violence, making women more vulnerable to violence. When the reasons for submissive behaviors towards violence are examined, it is stated that factors such as having children, low self-esteem, religious beliefs, social pressure, emotional attachment to a long-term relationship, running away from home, arranged marriage, being economically dependent on the spouse and low level of education are effective. Accepting violence encourages aggression and causes violent people to legitimize their actions. It is stated that submissive and accepting attitudes towards violence can be changed. Interventions aimed at empowering women play an important role in reducing attitudes accepting violence. It is anticipated that this project will create an opportunity for women to raise awareness about violence and change their accepting attitudes towards violence.

The proposed project consists of THREE stages. The first stage, PREPARATION stage; includes preparation of data collection tools, determination and informing of scholarship recipients, development of training content and tools, preliminary application and determination of the working group. The second stage is the IMPLEMENTATION stage, which includes collecting pre-test data, loading public transportation fees onto participants' cards for transportation, providing training to the intervention group, and collecting post-test data. The third stage is the MONITORING-EVALUATION stage, which is the stage of collecting follow-up test data and conducting analyses.

The research will be conducted as a randomized controlled parallel group intervention study. The universe of the research will consist of 7988 women registered in 24 Women's Education and Culture Centers (KEKM) affiliated with Altındağ Municipality. 1 center will be randomly selected from 24 Women's Education and Culture Centers for the sample of the research. In this study, the smallest sample size was determined as 43 for each group, totaling 86, at 80% statistical power and α=.05 significance level. Considering the 10% data loss in the determined sample size, it was planned to include a total of 94 participants, 47 for each group. The assignment of the women included in the research to the intervention (47 participants) and control (47 participants) groups will be done by randomization method. The aim is to implement the Laughter Yoga Supported Strong Woman, Safe Life Training Program face-to-face for an 8-week period for the participants in the intervention group. The 47 participants in the intervention group will be divided into 3 separate groups (16 participants, 16 participants and 15 participants) to increase interaction and experience sharing. The project team will implement the Laughter Yoga Supported Strong Woman, Safe Life Training Program consisting of 8 modules to 3 separate groups. The intervention group will be given a pre-test before the training, a post-test after the training and a follow-up test 1 month after the training is completed. It is planned to collect data by conducting a pre-test, post-test and follow-up test simultaneously with the experimental group without any intervention for the control group. Data will be collected using the Attitude Towards Violence in Close Relationships Scale, the Psychological Flexibility Scale and the Styles of Coping with Stress Scale. Institutional permission will be obtained from the Ankara University Ethics Committee and the Altındağ Municipality.

In this project, with the "Strong Woman, Safe Life Training Program Supported by Laughter Yoga", women will be provided with training on the Importance of Self-Knowledge and Communication, Stress and Coping Techniques, Gender, Empowerment

DETAILED DESCRIPTION:
The aim of this project is to examine the effects of the Laughter Yoga Supported Strong Woman, Safe Life Education Program applied to women on attitudes towards violence, stress coping styles and psychological flexibility.

The problem of violence against women is a public health problem that affects and concerns not only women at the individual level, but also children, all family members and therefore society. According to the data of the Turkish Statistical Institute in our country, 38% of women have been subjected to spousal or partner violence at some point in their lives. Violence or the threat of violence that causes fear, pain and anxiety in women from an individual perspective; constitutes an obstacle to women's more active and productive participation in economic and social life, especially in the private sphere. From a social perspective, the economic cost of violence against women is extremely high in terms of loss of working hours and wages, social services, legal and medical expenses.

Our country has a culturally patriarchal social structure. Living in a patriarchal order affects beliefs and attitudes towards the acceptance of violence, making women more vulnerable to violence. Living in a patriarchal order affects beliefs and attitudes towards acceptance of violence, making women more vulnerable to violence. When the reasons for submissive behaviors towards violence are examined, it is stated that factors such as having children, low self-esteem, religious beliefs, social pressure, emotional attachment to a long-term relationship, running away from home, arranged marriage, being economically dependent on the spouse and low level of education are effective. Accepting violence encourages aggression and causes violent people to legitimize their actions. It is stated that submissive and accepting attitudes towards violence can be changed. Interventions aimed at empowering women play an important role in reducing attitudes accepting violence. It is anticipated that this project will create an opportunity for women to raise awareness about violence and change their accepting attitudes towards violence.

The proposed project consists of THREE stages. The first stage, PREPARATION stage; includes preparation of data collection tools, determination and informing of scholarship recipients, development of training content and tools, preliminary application and determination of the working group. The second stage is the IMPLEMENTATION stage, which includes collecting pre-test data, loading public transportation fees onto participants' cards for transportation, providing training to the intervention group, and collecting post-test data. The third stage is the MONITORING-EVALUATION stage, which is the stage of collecting follow-up test data and conducting analyses.

The research will be conducted as a randomized controlled parallel group intervention study. The universe of the research will consist of 7988 women registered in 24 Women's Education and Culture Centers (KEKM) affiliated with Altındağ Municipality. 1 center will be randomly selected from 24 Women's Education and Culture Centers for the sample of the research. In this study, the smallest sample size was determined as 43 for each group, totaling 86, at 80% statistical power and α=.05 significance level. Considering the 10% data loss in the determined sample size, it was planned to include a total of 94 participants, 47 for each group. The assignment of the women included in the research to the intervention (47 participants) and control (47 participants) groups will be done by randomization method. The aim is to implement the Laughter Yoga Supported Strong Woman, Safe Life Training Program face-to-face for an 8-week period for the participants in the intervention group. The 47 participants in the intervention group will be divided into 3 separate groups (16 participants, 16 participants and 15 participants) to increase interaction and experience sharing. The project team will implement the Laughter Yoga Supported Strong Woman, Safe Life Training Program consisting of 8 modules to 3 separate groups. The intervention group will be given a pre-test before the training, a post-test after the training and a follow-up test 1 month after the training is completed. It is planned to collect data by conducting a pre-test, post-test and follow-up test simultaneously with the experimental group without any intervention for the control group. Data will be collected using the Attitude Towards Violence in Close Relationships Scale, the Psychological Flexibility Scale and the Styles of Coping with Stress Scale. Institutional permission will be obtained from the Ankara University Ethics Committee and the Altındağ Municipality.

In this project, with the "Strong Woman, Safe Life Training Program Supported by Laughter Yoga", women will be provided with training on the Importance of Self-Knowledge and Communication, Stress and Coping Techniques, Gender, Empowerment of Women, Violence and Its Effects on Women's Health, Non-Violent Communication, Combating Violence, and Psychological Health, thus contributing to the reduction of women's attitudes towards violence and their gaining a conscious attitude towards violence. The project's training program

ELIGIBILITY:
Inclusion Criteria Being a woman Being 18 years of age or older Having a partner, speaking, understanding Reading and writing in Turkish Being registered in a women's education and culture center

Exclusion Criteria Having any communication barrier Having a diagnosed psychiatric illness Having attended a planned training on violence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This project aims to empower women against intimate partner violence by providing training.
Enrollment: 1 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Attitudes Towards Violence in Close Relationships Scale | Within 3 months after the project starts
  It was planned to collect pre-test and post-test data from the intervention and control groups in a face-to-face environment using the Attitudes Towards Violence in Close Relationships Scale The "Attitudes Towards Violence in Close Relationships Scale-GGF"was adapted into Turkish by Toplu-Demirtaş et al. (2017). There are 17 items on the five-point Likert-type scale. As a result of the validity analyses, it was determined that the scale has three sub-dimensions as "abuse-8 items, Control-5 items and violence-4 items". In the instructions used, the participants were asked to rate how compatible each item was for them between 1 (Strongly Disagree) and 5 (Strongly Agree). Items 2, 4, 5, 8, 12, 13, 14 and 17 of the scale are reverse scored. Higher scores obtained from the scale reflect more accepting attitudes towards psychological and physical violence.
The Psychological Flexibility Scale | Within 3 months after the project starts
  It was planned to collect pre-test and post-test data from the intervention and control groups in a face-to-face environment using the Psychological Flexibility Scale. This measurement tool focuses on five different subcategories: Values and behavior in line with values (10 questions), being in the moment (7 questions), acceptance (5 questions), contextual self (3 questions), and separation (3 questions). Each question is subject to a scoring system between 1 and 7. This measurement tool was translated into Turkish by Karakuş and Akbay (2020). The 28 questions of the Psychological Flexibility Scale focus on five subcategories: Values and behavior in line with values, beingin the moment, acceptance,, contextual self and dissociation. Items 2, 3, 5, 6, 8, 18, 20, 22, 23, 24 and 25 are reverse scored. High scores obtained from each subcategory indicate high psychological flexibility.
The Ways of Coping with Stress Scale | Within 3 months after the project starts
  It was planned to collect pre-test and post-test data from the intervention and control groups in a face-to-face environment using the Ways of Coping with Stress Scale

IPD SHARING:
Plan to Share IPD: Undecided